CLINICAL TRIAL: NCT04822571
Title: Investigating the Reliability of Highly Dynamic 3D Motion Analysis Protocol in Adolescence and Adult Males
Acronym: CAM-FAI relia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S64417
Record Dates: First submitted 2021-03-16; First posted 2021-03-30 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Femoroacetabular Impingement
Keywords: 3D motion analysis; Reliability
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescent volunteers (Other): Adolescent males aged 12-16 years old
  Interventions: Other: Reliability of 3D motion analysis protocol
- Adult volunteers (Other): Adult males aged 25-35 years old
  Interventions: Other: Reliability of 3D motion analysis protocol

INTERVENTIONS:
Other: Reliability of 3D motion analysis protocol — The intrinsic and extrinsic reliability of the designed 3D motion analysis protocol is measured in cases of high velocity dynamic movement such as kicking a soccer ball.

SUMMARY:
Femoroacetabular impingement is an orthopedic condition that is primarily characterized by the presence of anatomic bony abnormalities in the femoral head and/or the acetabulum resulting in an abnormal contact between the two during hip motion, especially in positions of increased hip flexion and rotation, ultimately leading to hip pain.

The main study was initiated with the goal of exploring the etiology of FAI in a multidimensional and novel way that addresses the major gaps in literature. Within the main study a 3D motion capture protocol has been designed in line with the latest literature recommendations, which called for more hip ROM specific movements and athlete oriented 3D motion capture protocols that incorporate the spinopelvic complex. While the protocol surely contains movements that have been previously validated and published such as squats and lunges, a unique addition of high velocity soccer kicks and hop- lunges have been included.

Such additions elevate the relevancy of the 3D motion analysis protocol, however they also pose questions on how reliable and accurate these additions are. This is especially important a 3D motion analysis has a very subjective component, which is the placement of the skin markers by the clinician. Errors or alteration to markers placement between different sessions or different subjects have been shown to significantly affect the quality of data. Furthermore, not all physical movement can be properly documented using motion analysis. The velocity at which the movement is preformed combined with how complex it is can affect the quality of data collected by the motion analysis system. Also another important component is the uniqueness of the population recruited for the main study. Most studies with highly dynamic motion protocols have been validated and published on adult populations. Thus the investigators cannot use their findings liberally to compare with the adolescent protocol, as differences in patterns of motion between adults and adolescence have been documented. Indeed, a need to test the reliability of the investigators' protocol among their own study groups is highly imperative.

DETAILED DESCRIPTION:
Femoroacetabular impingement is an orthopedic condition that is primarily characterized by the presence of anatomic bony abnormalities in the femoral head and/or the acetabulum resulting in an abnormal contact between the two during hip motion, especially in positions of increased hip flexion and rotation, ultimately leading to hip pain. FAI can be radiologically classified into 3 types of morphology: Pincer, CAM and mixed type. Pincer morphology is mainly characterized on radiological films by an over-coverage of the acetabulum, has a high center edge angle and is seen in females more frequently. CAM morphology is characterized by an increase in bone formation at the femoral head-neck junction and is mainly identified by a large alpha angle on medical imaging scans. Unlike pincer, CAM morphology occurs mainly in males. Mixed morphology is a third type of FAI and consists of a combination of both CAM and pincer impingement characteristics. FAI has been increasingly garnering attention in the last two decades due to two main reasons.

The first reason is its recognition as a leading cause of hip pain in the young economically-active adult. Epidemiological reports show the average age of FAI patients is 28 years old. Furthermore, a significant number of FAI patients are athletes who have professional careers that heavily depend on their physical wellbeing. The second reason FAI has been in the spotlight of orthopedic research recently, is the growing evidence linking it to early cartilage and labral damage, and subsequently to the development of hip osteoarthritis (OA). Ganz and colleagues were the first to make this link and assumed that the presence of the inter-articular morphological abnormality leads to abutment of the femoral head-neck junction against the acetabular rim. This repeated mechanical abutment is assumed to then lead to acetabular labral damage and progressive breakdown of the chondrolabral junction, thereby leading to chondral defects and the eventual onset of OA. Hip OA by itself is an acknowledged source of pain/disability and is associated with an ever-increasing socioeconomic cost.

A recent systematic review on the prevalence of symptomatic hip morphology reported the prevalence of CAM type deformity to be 37%; the prevalence of pincer deformity was 67% in the general population. Interestingly, there was an almost 3:1 ratio of CAM deformity in an athletic population compared with non-athletes. This was not the case for pincer deformity. Furthermore, such morphological findings are increasingly being reported in the adolescent athletic population specifically. A number of recent studies found a markedly higher prevalence of cam deformities in asymptomatic adolescents participating in, specifically, soccer, ice-hockey and basketball as compared with their non-athlete controls. Such reports have led researchers to speculate whether participating in high intensity physical activity at the critical period of bone maturation prior to femoral physis closure (10 - 15 years of age) could cause CAM deformity post femoral physis closure (15 -18 years of age old). It is hypothesized that a CAM in this population could form either due to new bone formation at the anterosuperior head-neck junction, or be induced by changes in the shape of the growth plate due to high shear forces acting on the growing hip during these athletic activities. However, as of date there is no concrete evidence to support this hypothesis. Consequently, the reasons behind the formations of CAM deformity in adolescent athletes remain unclear and call for further research. Such research is imperative to increase our understanding of the effect high training load can have on the wellbeing and long term health of young athletes.

It is with this background in mind that the main study was initiated with the goal of exploring the etiology of FAI in a multidimensional and novel way that addresses the major gaps in literature. Within the main study a 3D motion capture protocol has been designed in line with the latest literature recommendations, which called for more hip ROM specific movements and athlete oriented 3D motion capture protocols that incorporate the spinopelvic complex. While the protocol surely contains movements that have been previously validated and published such as squats and lunges, a unique addition of high velocity soccer kicks and hop- lunges have been included.

Such additions elevate the relevancy of the 3D motion analysis protocol, however they also pose questions on how reliable and accurate these additions are. This is especially important a 3D motion analysis has a very subjective component, which is the placement of the skin markers by the clinician. Errors or alteration to markers placement between different sessions or different subjects have been shown to significantly affect the quality of data. Furthermore, not all physical movement can be properly documented using motion analysis. The velocity at which the movement is preformed combined with how complex it is can affect the quality of data collected by the motion analysis system. Also another important component is the uniqueness of the population recruited for the main study. Most studies with highly dynamic motion protocols have been validated and published on adult populations. Thus the investigators cannot use their findings liberally to compare with the adolescent protocol, as differences in patterns of motion between adults and adolescence have been documented. Indeed, a need to test the reliability of the investigators' protocol among their own study groups is highly imperative.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: adolescent males aged 12-16 years old
* Group 2: adult males aged 25-35 years old

Exclusion Criteria:

- Volunteers who received major prior surgery of the lower limbs or with any pathology, injury or disorder known to affect the locomotor system

Ages: 12 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Kinematic parameters in order for reliability | within a time interval of 1 month
  The construction of all kinematic measurements in order for reliability using 3D motion analysis

SECONDARY OUTCOMES:
Copenhagen Hip and Groin Outcome Score (HAGOS) | within a time interval of 1 month
  The assessment of symptoms, activity limitations, participation restrictions and QOL in physically active, young to middle-aged patients with long-standing hip and/or groin pain
International Hip Outcome Tool (IHOT) | within a time interval of 1 month
  To obtain subjective measures of symptoms, as well as determining emotional and social health status

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Ghijselings, M.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No